CLINICAL TRIAL: NCT00344708
Title: Transplantation of Tissue Cultured Human Amniotic Epithelial Cells Onto Damaged Ocular Surfaces
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Potential subjects did not meet eligibility criteria
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, James McCulley, Chairman - Department of Ophthalmology, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0399-090
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Corneal Epithelial Dystrophy
Keywords: Tissue-Cultured Human Amniotic Epithelial Cells onto damaged corneal surface

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Transplantation of Tissue-Cultured Human Amniotic Epithelial Cells

SUMMARY:
To investigate the effect of using tissue cultured human amniotic epithelial cells to re-establish severely damaged ocular surfaces. Specifically, to determine the efficacy of transplanted tissue cultured amniotic epithelial cells on persistent corneal epithelial defect, a potential visual threaten ocular disorder.

DETAILED DESCRIPTION:
Ocular surface diseases and injury caused by chemicals, result in chronic ulceration, and may never be able to be healed normally, and may lead to permanent vision loss. Standard medical treatments often fail. Histologically and somehow functionally, human amniotic cells are similar to ocular surface cells, and these cells have been shown to be safe to be transplanted to another subject and will not be rejected by the recipient. In animal studies, amniotic cells demonstrated that they can re-establish the integrity of ocular surface in more than 30% of recipients without apparent toxic side effects. This study will investigate this novel strategy for its effect on human ocular surface disorder. It will provide a potential alternative therapy for this difficult and devastating disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with corneal epithelial defects and ulcers that have persisted for 4 weeks or longer, regardless of their cause. These patients will have received traditional medical therapy, including correcting the underlying causes, suppressing inflammation, and augmenting the tissue healing processes, but the epithelial defects have persisted.

Exclusion Criteria:

* Patients who are pregnant or under age 18 will be excluded.
* Placentas will not be used if the following problems are present:

  * If the mother has an infection at the time of her baby's birth;
  * If the mother has a high risk of developing infection due to intravenous drug use or other factors;
  * If the mother has diabetes, arthritis, or raised blood pressure;
  * If the baby is unhealthy;
  * If there is evidence of infection of the womb (uterus) and afterbirth (placenta) at the time of delivery.

Ages: 18 Years to 88 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2000-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Ocular surface healing | 30 days following initiation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: James P. McCulley, M.D., Principal Investigator — University of Texas, Southwestern Medical Center at Dallas
Locations (2):
- United States (2):
  - Aston Ambulatory Care Center, Dallas, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas